CLINICAL TRIAL: NCT02027090
Title: High Dose Versus Routine Dose Icotinib in Pretreated Non-small Cell Lung Cancer Patients With Stable Disease: a Phase II Randomized Study
Brief Title: High Dose Versus Routine Dose Icotinib in Advanced Non-small Cell Lung Cancer Patients With Stable Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV17
Record Dates: First submitted 2014-01-01; First posted 2014-01-03 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Higher dose icotinib (Experimental): Patients with stable disease after 8-week routine dose icotinib treatment, are randomly assigned to higher dose icotinib group to receive icotinib with a dose of 375 mg three times per day, till progressive disease or unaccepted toxicity.
  Interventions: Drug: Higher dose icotinib
- Routine dose icotinib (Active Comparator): Patients with stable disease after 8-week routine dose icotinib treatment, are administered with icotinib with a dose of 125 mg three times per day, till progressive disease or unaccepted toxicity.
  Interventions: Drug: Routine dose icotinib

INTERVENTIONS:
Drug: Routine dose icotinib — Icotinib is administered 125 mg three times daily.
  Other Names: Commana
  Arms: Routine dose icotinib
Drug: Higher dose icotinib — After 8-week induction of icotinib with a dose of 125 mg three times daily, icotinib is administered 375 mg three times per day.
  Other Names: Commana
  Arms: Higher dose icotinib

SUMMARY:
We hypothesize that higher dose icotinib is related with better efficacy. The primary objective is to compare the progression-free survival of higher dose and routine dose of icotinib in treating pretreated advanced non-small cell lung cancer patients with stable disease after 8-week routine dose icotinib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB/IV lung cancer(exclude patients confirmed by sputum cytology);
* Pretreated with at least 1 platinum-based chemotherapy;
* No previous targeted treatment such as gefitinib, erlotinib;
* With a measurable disease(longest diameters >=10mm with Spiral computed tomography (CT)and >=20mm with conventional CT) according to RECIST Criteria;
* WHO performance status(PS)<= 2;
* Adequate organ functions;
* Signed and dated informed consent before the start of specific protocol procedures.

Exclusion Criteria:

* Allergic to icotinib;
* Patients with metastatic brain tumors with symptoms;
* Experience of Anti-EGFR(the epidermal growth factor receptor) Monoclonal Antibody or small molecular compounds therapy such as gefitinib, erlotinib or Cetuximab;
* Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 5 months

SECONDARY OUTCOMES:
Overall survival | 18 months
Response rate assessed using the RECIST criteria | 2 months
The number of patients who suffered adverse events | 30 months
  Adverse events are assessed by Common Terminology Criteria for Adverse Events v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital Affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China